CLINICAL TRIAL: NCT02905071
Title: Study of the Psychometric Properties of the Scale of Well-being at Work: The Serenat Study
Brief Title: Validation of a Scale of Well-being at Work
Acronym: SERENAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2012_63; 2013-A00831-44 (Other: ID-RDB number, ANSM)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2018-11

CONDITIONS: Adjustment Disorder
Keywords: mental health; well-being at work; screening; psychosocial risk; psychometrics; questionnaire; job stress
MeSH Terms: conditions — Adjustment Disorders; Psychological Well-Being; Occupational Stress | interventions — BaseLine dental cement; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study 1 Group 1 G1 (n =50) (Experimental): filling of Serenat at baseline (T1)
  Interventions: Other: filling of Serenat at baseline (T1)
- Study 1 Group 2 G2 (n=50) (Experimental): Serenat at baseline T1 and 3 others questionnaires
  Interventions: Other: Serenat at baseline T1 and 3 others questionnaires
- Study 1 Group 3 G3 (n =50) (Experimental): filling of Serenat at baseline T1 and T2 (one week after baseline).
  Interventions: Other: filling of Serenat, HADS, STAY-Y and BDI at baseline T1
- Study 2 Ancillary study (n=50) (Experimental): filling of Serenat, HADS, STAY-Y and BDI at baseline T1
  Interventions: Other: Serenat at baseline T1 and 3 others questionnaires

INTERVENTIONS:
Other: filling of Serenat at baseline (T1) — Patients who consult occupational doctor complete the serenat questionnaire.The time taken to complete the serenat scale is about 5 minutes.
  Other Names: filling of Serenat at T1 (baseline)
  Arms: Study 1 Group 1 G1 (n =50)
Other: Serenat at baseline T1 and 3 others questionnaires — Subjects who consult occupational doctor complete the 4 questionnaires.The time taken to complete the 4 questionnaires is about 15 minutes.
  Other Names: Serenat and 3 others questionnaires at T1
  Arms: Study 1 Group 2 G2 (n=50); Study 2 Ancillary study (n=50)
Other: filling of Serenat, HADS, STAY-Y and BDI at baseline T1 — Patients who consult a psychiatrist in a stress anxiety unit complete the 4 questionnaires.
  Other Names: filling of Serenat at baseline T1 and T2 (one week later)
  Arms: Study 1 Group 3 G3 (n =50)

SUMMARY:
The main objective of this work is to explore the psychometric properties of scale of well-being at work called "Serenat" in order to validate it. Secondary objectives are to study the influence of socio-demographic characteristics of the subjects on the results of Serenat and to describe the results on subjects monitored among an adult psychiatric population.

DETAILED DESCRIPTION:
This is a cross sectional survey. 200 subjects were selected among people having consulted an occupational doctor to validate the scale in the general population (study 1), and 50 subjects among a psychiatric population for the ancillary study (study 2).

The Serenat Scale is a self-report questionnaire composed of 20 items. All items are scored on a four point Likert scale ranging from 0 (strongly disagree) to 3 (strongly agree) resulting in a range of 0 to 60. The 20 items are related to different domains. 10 items explore psychological balance at work: relaxation (item 1), sleep quality (item 2), concentration (item 3), form (item 4), sense of security (item 5), satisfaction (item 6), quality of relationships and contacts at work (item 7), voltage or aggressiveness (item 8), optimism for the future from a professional point of view (item 9), life balance (item 10). 10 items are related to working conditions and organization of work: comfort of the working environment (item 11), time constraint (item 12), sense of competence (item 13), decision latitude (item 14), interest at work and variety of tasks (item 15), recognition (item 16), professional support (item 17), communication and transfer of information (item 18), human conflict (item 19), satisfactory work schedules (item 20).

ELIGIBILITY:
Inclusion Criteria:

* agree to participate, exert a professional activity for at least 3 months at the time of inclusion, consult an occupational doctor or go to consultations related to stress and anxiety, read and be able to respond to the scale,

Exclusion Criteria:

* not be acting on work stoppage, nor pregnant, be capable of consent, not benefit from any legal protection regime and not be deprived of freedom.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Serenat scale | At baseline (T1)
  For Group 1, Group 2, Group 3: The Serenat Scale is a self-report questionnaire composed of 20 items. All items are scored on a four point Likert scale ranging from 0 (strongly disagree) to 3 (strongly agree) resulting in a range of 0 to 60. The 20 items are related to different domains. 10 items explore psychological balance at work. 10 items are related to working conditions and organization of work.

SECONDARY OUTCOMES:
Serenat scale | one week after baseline (T2)
  For Group 3: The Serenat Scale is a self-report questionnaire composed of 20 items. All items are scored on a four point Likert scale ranging from 0 (strongly disagree) to 3 (strongly agree) resulting in a range of 0 to 60. The 20 items are related to different domains. 10 items explore psychological balance at work. 10 items are related to working conditions and organization of work.
Hospital Anxiety and Depression Scale (HADS) | At baseline (T1)
  For group 2: The scale allows to detect anxiety and depression using 14 items rated from 0-3.
State-Trait Anxiety inventory (STAI-Y) | At baseline (T1)
  For Group: Self-administered questionnaire of 20 items side on 4 levels from 'not at all' to one side "many" side 4 (total score of 20-80). It measures an intensity of more anxiety and is not related to an anxiety disorder
The Beck depression inventory (BDI-21) | At baseline (T1)
  For Group, Self-assessment questionnaire measuring the severity of depression

CONTACTS AND LOCATIONS:
Overall Officials: Dominique SERVANT, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Fontan 2, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andrea H, Bultmann U, Beurskens AJ, Swaen GM, van Schayck CP, Kant IJ. Anxiety and depression in the working population using the HAD Scale--psychometrics, prevalence and relationships with psychosocial work characteristics. Soc Psychiatry Psychiatr Epidemiol. 2004 Aug;39(8):637-46. doi: 10.1007/s00127-004-0797-6. PMID 15300374
- [Background] Stansfeld S, Candy B. Psychosocial work environment and mental health--a meta-analytic review. Scand J Work Environ Health. 2006 Dec;32(6):443-62. doi: 10.5271/sjweh.1050. PMID 17173201
- [Background] Melchior M, Caspi A, Milne BJ, Danese A, Poulton R, Moffitt TE. Work stress precipitates depression and anxiety in young, working women and men. Psychol Med. 2007 Aug;37(8):1119-29. doi: 10.1017/S0033291707000414. Epub 2007 Apr 4. PMID 17407618
- [Result] Servant D, Drumez E, Raynal S, Demarty AL, Salembier A, Deschepper MH, Bizet MA, Pisanu-Zimny A, Culem JB, Labreuche J, Duhamel A, Vaiva G. [Elaboration and psychometric properties of a well-being scale at work. The Serenat study among employees in occupational medicine unit]. Rev Epidemiol Sante Publique. 2019 Sep;67(5):303-309. doi: 10.1016/j.respe.2019.05.011. Epub 2019 Jun 28. French. PMID 31262608